CLINICAL TRIAL: NCT04741789
Title: Managed Access Program (MAP) Cohort Treatment Plan CINC280A02001M to Provide Access to Capmatinib, for MET Exon 14 Skipping Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Treatment Plan CINC280A02001M to Provide Access to Capmatinib, for MET Exon 14 Skipping Non-Small Cell Lung Cancer (NSCLC)
Status: Available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CINC280A02001M
Record Dates: First submitted 2021-02-03; First posted 2021-02-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small Cell Lung; Non-Small Cell Lung Cancer; Non-Small-Cell Lung Carcinoma; Nonsmall Cell Lung Cancer
Keywords: Non-small cell lung carcinoma; NSCLC; Treatment of lung cancer; Lung cancer; Lung adenocarcinoma; Squamous cell lung carcinoma; Large-cell lung carcinoma; Non small cell lung carcinoma; Non small cell lung cancer; Non-small cell lung cancer; Large cell lung carcinoma; Large cell lung cancer; MET Exon 14 skipping; skipping; Exon 14
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma of Lung | interventions — capmatinib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Capmatinib — Tablet for oral use, dose Up to 400mg, twice daily
  Other Names: INC280

SUMMARY:
The purpose of this Managed Access Program (MAP) Cohort Treatment Plan is to provide guidance to the Physician for the treatment and monitoring of patients in the Cohort MAP.

The Physician should follow the suggested treatment guidelines. Furthermore, the Physician must comply with the MAP Agreement Letter and applicable local laws and regulations.

DETAILED DESCRIPTION:
Prior to inclusion of a patient in the Cohort, the requesting Physician must submit a request for access to the product in GEMS (Grants, External Requests and Managed Access System) accessible through https://www.novartis.com/our-focus/healthcare-professionals/managedaccess- programs providing the rationale for the request and relevant medical history of the patient. The request is then assessed against the MAP and Cohort inclusion/exclusion criteria by the medical team experienced with the product and indication. Upon the required approvals, the patient is included in the Cohort.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this Treatment Plan have to meet all of the following criteria:

1. Age ≥ 18 years
2. Patients with advanced or metastatic MET exon 14 skipping (METex14) NSCLC. In European Union countries: Patients with advanced or metastatic MET exon 14 skipping (METex14) NSCLC who have received a prior line of therapy.
3. Patients must have adequate organ function including the following laboratory values at the program enrollment:

   * Calculated creatinine clearance (using Cockcroft-Gault formula) ≥ 45 mL/min
   * Total bilirubin ≤ 1.5 x ULN
   * Aspartate transaminase (AST) ≤ 3 x ULN, except for patients with liver metastasis, who may only be included if AST ≤ 5 x ULN
   * Alanine transaminase (ALT) ≤ 3 x ULN, except for patients with liver metastasis, who may only be included if ALT ≤ 5 x ULN
   * Alkaline phosphatase (ALP) ≤ 5.0 x ULN
   * Asymptomatic serum amylase ≤ grade 2. Patients with grade 1 or grade 2 serum amylase at the beginning of the treatment must be confirmed to have no signs and/or symptoms suggesting pancreatitis or pancreatic injury (e.g., elevated P-amylase, abnormal imaging findings of pancreas, etc.)
   * Serum lipase ≤ ULN
4. Written patient informed consent must be obtained prior to start of treatment in accordance with local laws and regulations.

Exclusion Criteria :

Patients eligible for this Treatment Plan must not meet any of the following criteria:

1. Participants with known hypersensitivity to any of the excipients of Capmatinib (crospovidone, mannitol, microcrystalline cellulose, povidone, sodium lauryl sulfate, magnesium stearate, colloidal silicon dioxide, and various coating premixes).
2. Presence or history of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention).
3. Thoracic radiotherapy to lung fields ≤ 4 weeks prior to starting Capmatinib or patients who have not recovered from radiotherapy-related toxicities. For all other anatomic sites (including radiotherapy to thoracic vertebrae and ribs), radiotherapy ≤ 2 weeks prior to starting Capmatinib or patients who have not recovered from radiotherapy-related toxicities. Palliative radiotherapy for bone lesions ≤ 2 weeks prior to starting Capmatinib is allowed.
4. Major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) within 4 weeks prior (2 weeks for resection of brain metastases) to starting Capmatinib or who have not recovered from side effects of such procedure. Video-assisted thoracic surgery (VATS) and mediastinoscopy will not be counted as major surgery and patients can be enrolled in the program ≥ 1 week after the procedure
5. Patients receiving treatment with strong inducers of CYP3A4 that cannot be discontinued at least 1 week prior to the start of treatment with Capmatinib and for the duration of the treatment
6. Impairment of GI function or GI disease that may significantly alter the absorption of Capmatinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome)
7. Unable or unwilling to swallow tablets as per dosing schedule
8. Patients receiving treatment with any enzyme-inducing anticonvulsant that cannot be discontinued at least 1 week before first dose of Capmatinib, and for the duration of the treatment. Patients on non-enzyme-inducing anticonvulsants are eligible
9. Other severe, acute, or chronic medical or psychiatric conditions, substance abuse or laboratory abnormalities that in the opinion of the treating physician may increase the risk associated with the treatment,
10. Any other condition that would, in the treating physician's judgment, contraindicate treatment due to safety concerns e.g., active infection (including active hepatitis B and C, SARS-CoV-2), inflammation, intestinal obstruction, unable to swallow medication, social/ psychological issues, etc.
11. Participants who received live vaccines (e.g., intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella, TY21a typhoid vaccines and COVID 19 vaccines) within 30 days prior to the first dose of study treatment.
12. Pregnant or nursing (lactating) women
13. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 7 days after stopping treatment. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) total hysterectomy, or tubal ligation at least six weeks before taking treatment. In case of unilateral oophorectomy, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female subjects on the program the vasectomized male partner should be the sole partner for that subject
    * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking treatment.

    Note: Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before program entry. In the case of unilateral oophorectomy, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
14. Sexually active males unless they use a condom during intercourse while taking drug and for 7 days after stopping treatment and should not father a child in this period. A condom is required for all sexually active males to prevent them from fathering a child AND to prevent delivery of capmatininb via seminal fluid to partner. In addition, male participants must not donate sperm for the time period specified above

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult